CLINICAL TRIAL: NCT04724759
Title: The Effect of Opioid-Free Anesthesia in TMJ Surgery: A Prospective Study
Brief Title: The Effect of Opioid-Free Anesthesia in TMJ Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jingping Wang, MD, Ph.D., Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020P003873
Record Dates: First submitted 2020-12-30; First posted 2021-01-26 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Opioid
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Dexmedetomidine; Ketamine; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Opioid-free Anesthesia (Experimental): Patients in this arm will not receiving opioids but the total intravenous anesthetic during surgery. Patients in this group will receive an infusion of lidocaine, ketamine, or dexmedetomidine supplemented with other intravenous analgesics and intravenous and inhaled anesthetics.
  Interventions: Drug: Dexmedetomidine / Ketamine / Lidocaine
- Standard Anesthesia (No Intervention): Patients in this arm will undergo the standard of care and receive opioids as part of their anesthetic regimen.

INTERVENTIONS:
Drug: Dexmedetomidine / Ketamine / Lidocaine — Patients in this group will receive an infusion of lidocaine, ketamine, or dexmedetomidine supplemented with other intravenous analgesics and intravenous and inhaled anesthetics, as needed clinically. This includes administration of 5 mcg/kg/min of ketamine plus 0.5 - 1.0 µg/kg/hr of dexmedetomidine (Precedex) as a continuous infusion, started from induction to stop one hour before surgery is anticipated to end.
  Other Names: Precedex
  Arms: Opioid-free Anesthesia

SUMMARY:
This study aims is to evaluate the effect of opioid free total intravenous anesthesia on postoperative quality of recovery in patients undergoing oral and maxillofacial surgery (OMF) temporomandibular joint (TMJ) surgery.

DETAILED DESCRIPTION:
This study will enroll 60 patients undergoing TMJ surgery at Massachusetts General Hospital. Anesthetic care will be standardized according to current institutional standards of care. Intraoperative clinicians will not be blinded to group assignment. Patients will be randomized to one of two groups:

* Group 1 - Opioid-free Anesthesia Patients: Patients who are not receiving opioids but the total intravenous anesthetic during surgery.
* Group 2 - Standard Anesthesia Patients: Patients who undergo the standard of care and receive opioids as part of their anesthetic regimen.

Both groups employ strategies that are routinely used as part of standard clinical practice for TMJ surgery. Patients will otherwise receive the institutional standards of care for their surgical procedure and perioperative care.

Following intraoperative drug administration patients will be followed until discharge from the PACU to assess study endpoints while in the hospital. At the time of discharge from the PACU, members of the study team will ask the patient to compete a brief survey on their satisfaction with pain management.

Patients in this study will be anticipated to be discharged the same day as the surgical procedure. At the time of hospital or PACU discharge, the patient will be provided with a Medication Diary. This will be used to record pain medication administration in the first 48 hours after surgery, as well as any pain or complication they might experience at home.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 (inclusive)
* Scheduled for TMJ surgery (including both unilateral and bilateral procedures)
* Planned arthroscopic surgical procedure
* Preoperative plan to discharge the same day

Exclusion Criteria:

* Inability to provide written informed consent
* Pregnant patients
* Open TMJ Surgeries
* Planned overnight admission
* Mental status disorder or patient who are unable to communicate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2023-04-23 (Actual); Study Completion 2023-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jingping Wang, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Opioid-free Anesthesia | Standard Anesthesia
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid-free Anesthesia | Standard Anesthesia | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 1 | 1 | 2
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38.0 [26.0 to 51.8] | 36.0 [27.5 to 53.3] | 37.50 [26.00 to 52.50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 53
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 24 | 25 | 49
  Unknown or Not Reported | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 23 | 24 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: Pain will be measured using the eleven point (0 to 10) numeric rating scale with higher values representing a worse outcome. Pain scores will be recorded every 15 minutes until discharge from the post-anesthesia care unit (PACU) and at 12 and 24 hours postoperatively. Clinically documented pain scores will be recorded. Our primary outcome will be the worst documented pain score while in the PACU. Additional pain score time points will be evaluated as secondary endpoints.
Time Frame: Through in-hospital study completion, an average of 1 day
Population: Worst PACU Pain Score - Opioid Free 4.9 (2.4)
  Worst PACU Pain Score - Standard of Care (Control) 4.4 (2.8)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Opioid-free Anesthesia | Standard Anesthesia
Number analyzed (Participants) | 30 | 30
units on a scale | 4.9 (2.4) | 4.4 (2.8)

2. Secondary Outcome: Perioperative Opioid Use
Description: Intraoperative and postoperative opioid consumption in the first 12, 24 and 48 hours postoperatively will be evaluated.
Time Frame: 48 hours postoperatively
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Opioid-free Anesthesia | Standard Anesthesia
Number analyzed (Participants) | 30 | 30
morphine milligram equivalents | 21 (70) | 20 (66.7)

3. Secondary Outcome: Rescue Analgesia in the PACU
Description: Use, dosage and time to use of rescue analgesia in the PACU will be reported.
Time Frame: Through in-hospital study completion, an average of 1 day
Population: Time to Rescue Analgesia (minutes), Median [Q1,Q3] Opioid Free: 104.0 [84.5, 224.0] Standard of Care (Control): 83.5 [51.1, 155.0]
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Opioid-free Anesthesia | Standard Anesthesia
Number analyzed (Participants) | 30 | 30
Minutes | 104.0 [84.5 to 224.0] | 83.5 [51.1 to 155.0]

4. Secondary Outcome: Pain Satisfaction
Description: Self-report pain satisfaction will be assessed at the time of PACU discharge using the Revised American Pain Society Patient Outcome Questionnaire.
  This survey asked patients to grade pain either the pain experienced (graded from a 0-10 scale, 0 bring no pain and 10 being the worst pain possible), pain associated with certain movements (0-10 scale, 0 does not interfere and 10 being completely interferes), pain associated with emotions (0-10 scale, 0 not at all and 10 being extremely), side effects (0-10 scale, 0 none and 10 Severe), pain relief (0-10 scale, 0 no relief and 10 being complete relief), and satisfaction (0-10 scale, 0 extremely dissatisfied and 10 being extremely satisfied).
Time Frame: Completed upon the patient reaching PACU Phase I in the hospital, up to approximately 6 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid-free Anesthesia | Standard Anesthesia
Number analyzed (Participants) | 30 | 30
Participants
  0 | 1 | 0
  1 | 1 | 0
  2 | 0 | 0
  3 | 0 | 1
  4 | 0 | 0
  5 | 1 | 1
  6 | 0 | 0
  7 | 0 | 1
  8 | 5 | 6
  9 | 2 | 2
  10 | 18 | 14
  No Survey Completed | 2 | 5

5. Secondary Outcome: Incidence of Opioid Related Adverse Effects
Description: The incidence of ileus, nausea/vomiting, and pruritis will be reported.
Time Frame: 48 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid-free Anesthesia | Standard Anesthesia
Number analyzed (Participants) | 30 | 30
Participants | 6 | 14

6. Secondary Outcome: Length of Stay (PACU Discharge)
Description: Length of PACU and hospital stay will be reported.
Time Frame: Through in-hospital study completion, an average of 1 day
Measure: Median (Inter-Quartile Range); unit: minutes for PACU
Arm/Group | Opioid-free Anesthesia | Standard Anesthesia
Number analyzed (Participants) | 30 | 30
minutes for PACU | 227.0 [192.5 to 268.0] | 206.0 [176.3 to 244.8]

7. Secondary Outcome: Percocet Use
Description: The total dose of Percocet used at 24 and 48 hours after surgery will be reported.
Time Frame: 48 hours postoperatively
Population: Postoperative Percocet Use (mg) Opioid Free: 0 [0, 25] Standard of Care (Control): 5 [0, 25]
Measure: Median (Inter-Quartile Range); unit: Milligrams
Arm/Group | Opioid-free Anesthesia | Standard Anesthesia
Number analyzed (Participants) | 30 | 30
Milligrams | 0 [0 to 25] | 5 [0 to 25]

8. Secondary Outcome: Length of Stay (Hospital Discharge)
Description: Time to Hospital Discharge will be reported.
Time Frame: Through in-hospital study completion, an average of 1 day
Measure: Median (Inter-Quartile Range); unit: Time to Hospital Discharge (hours)
Arm/Group | Opioid-free Anesthesia | Standard Anesthesia
Number analyzed (Participants) | 30 | 30
Time to Hospital Discharge (hours) | 4.1 [3.4 to 4.8] | 3.8 [3.0 to 4.3]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the trial. Each participant was assessed within the 48 hours after their scheduled surgery.
Arm/Group | Opioid-free Anesthesia | Standard Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 9/30 | 18/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Opioid-free Anesthesia (N=30) | Standard Anesthesia (N=30)
Nausea (Gastrointestinal disorders) | 5 | 9
Itching Sensation (Skin and subcutaneous tissue disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1
Intestinal/Bowel Obstruction (Gastrointestinal disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT04724759/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT04724759/ICF_001.pdf